CLINICAL TRIAL: NCT02685605
Title: A Multicenter Randomized Phase III Trial on INTraoperative RAdiotherapy in Newly Diagnosed GliOblastoma Multiforme (INTRAGO II)
Brief Title: Intraoperative Radiotherapy in Newly Diagnosed Glioblastoma Multiforme
Acronym: INTRAGO-II
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Carl Zeiss Meditec AG (Industry); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Frank A. Giordano, PI (Chair), Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTRAGO-II; ARO-2016-1 (Other: Working Party for Radiation Oncology (ARO) of the DKG); AG-NRO-03 (Other: German Society for Radiation Oncology (DEGRO))
Record Dates: First submitted 2016-02-05; First posted 2016-02-19 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Intraoperative Radiotherapy; Radiotherapy Dose Escalation
MeSH Terms: conditions — Glioblastoma | interventions — Chemoradiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Experimental Arm (A) (Experimental): Standard surgery plus intraoperative radiotherapy (20-30 Gy) followed by radiochemotherapy (EBRT: 60 Gy, 75 mg/m2/d temozolomide) and adjuvant chemotherapy with 150-200 mg/m2/d temozolomide per cycle (5/28 days).
  Interventions: Procedure: Standard surgery; Radiation: Intraoperative radiotherapy; Radiation: Radiochemotherapy; Drug: Temozolomide
- Control Arm (B) (Active Comparator): Standard surgery followed by radiochemotherapy (EBRT: 60 Gy, 75 mg/m2/d temozolomide) and adjuvant chemotherapy with 150-200 mg/m2/d temozolomide per cycle (5/28 days).
  Interventions: Procedure: Standard surgery; Radiation: Radiochemotherapy; Drug: Temozolomide

INTERVENTIONS:
Procedure: Standard surgery
Radiation: Intraoperative radiotherapy — Dose to applicator surface: 20-30 Gy; Carl Zeiss INTRABEAM System. IORT with a surface dose of 30 Gy is recommended.Should the proximity to any risk structure not allow to apply 30 Gy, a dose reduction by up to 10 Gy (resulting in a surface dose of 20 Gy) is allowed.
  Other Names: IORT
  Arms: Experimental Arm (A)
Radiation: Radiochemotherapy — EBRT to 60 Gy plus 75 mg/m2/d temozolomide
Drug: Temozolomide — Adjuvant chemotherapy with 150-200 mg/m2/d temozolomide per cycle (5/28 days).

SUMMARY:
INTRAGO II resembles a multicentric, prospective, randomized, 2-arm, open-label clinical phase III trial which tests if the median progression-free survival (PFS) of patients with newly diagnosed glioblastoma multiforme (GBM) can be improved by the addition of intraoperative radiotherapy (IORT) to standard radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 and ≤ 80 years
2. Karnofsky Performance Score (KPS) ≥ 60%
3. Supratentorial T1-Gd enhancing lesion(s) amenable to total resection
4. Legal capacity and ability of subject to understand character and individual consequences of the clinical trial
5. Patient's written IC obtained at least 24h prior to surgery
6. For women with childbearing potential: adequate contraception
7. Patients must have adequate organ functions

   Bone marrow function:
   * Platelets ≥ 75.000/μL
   * WBC ≥ 3.000/μL
   * Hemoglobin ≥ 10.0 g/dL

   Liver Function:
   * ASAT and ALAT ≤ 3.0 times ULN
   * ALP ≤ 2.5 times ULN
   * Total Serum Bilirubin < 1.5 times ULN

   Renal Function:
   * Serum Creatinine ≤ 1.5 times ULN

   Inclusion Criteria Related to Surgery:
8. IORT must be technically feasible
9. Histology supports diagnosis of GBM

Exclusion Criteria

1. Multicentric disease (e.g. in both hemispheres) or non-resectable satellite lesions
2. Previous cranial radiation therapy
3. Cytostatic therapy / chemotherapy for cancer within the past 5 years
4. History of cancers or other comorbidities that limit life expectancy to less than five years
5. Previous therapy with anti-angiogenic substances (such as bevacizumab)
6. Technical impossibility to use MRI or known allergies against MRI and/or CT contrast agents
7. Participation in other clinical trials testing cancer-derived investigational agents/procedures.
8. Pregnant or breast feeding patients
9. Fertile patients refusing to use safe contraceptive methods during the study

   Exclusion Criteria Related to Surgery:
10. Active egress of fluids from a ventricular defect
11. In-field risk organs and/or IORT dose >8 Gy to any risk organ

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival | 24 Months
  Determined according to modified Response Assessment in Neuro-Oncology (RANO) criteria and serial perfusion imaging

SECONDARY OUTCOMES:
Median Overall Survival | 24 Months
PFS within a 1-2 cm margin around the cavity | 24 Months
  Determined by serial contrast-enhanced MRI scans using modified RANO criteria and serial perfusion imaging
OS with respect to Age | 24 Months
  Median overall survival of patients <65 vs. ≥ 65 years
PFS with respect to Age | 24 Months
  Progression-free survival of patients <65 vs. ≥ 65 years; determined according to modified RANO criteria and serial perfusion imaging
OS with respect to KPS | 24 Months
  Median overall survival of patients with KPS 80-100% vs. 60-70%
PFS with respect to KPS | 24 Months
  Progression-free survival of patients with KPS 80-100% vs. 60-70%; determined according to modified RANO criteria and serial perfusion imaging
OS with respect to thickness of anticipated T1-Gd-enhancing (remaining) tumor margin | 24 Months
  Thickness of anticipated T1-Gd-enhancing (remaining) tumor margin as per the discretion of the surgeon (margin ≥0.5 cm or multiple spots of residual tumor within the cavity vs. <0.5 cm)
PFS with respect to thickness of anticipated T1-Gd-enhancing (remaining) tumor margin | 24 Months
  Thickness of anticipated T1-Gd-enhancing (remaining) tumor margin as per the discretion of the surgeon (margin ≥0.5 cm or multiple spots of residual tumor within the cavity vs. <0.5 cm); determined according to modified RANO criteria and serial perfusion imaging
OS with respect to extent of resection | 24 Months
  Early postoperative MRI scans must be used to determine the extent of resection (EoR). The EoR is given as sum of all maximum diameters of residual lesions in cm. OS will be calculated for the following groups:
  * Max Diameter group 0: 0 cm (no residual tumor)
  * Max Diameter group 1: >0 to ≤1.5 cm (cumulative if multiple residual lesions)
  * Max Diameter group 2: >1.5 cm (cumulative if multiple residual lesions)
PFS with respect to extent of resection | 24 Months
  Early postoperative MRI scans must be used to determine the extent of resection (EoR). The EoR is given as sum of all maximum diameters of residual lesions in cm. PFS will be determined according to modified RANO criteria and serial perfusion imaging for the following groups:
  * Max Diameter group 0: 0 cm (no residual tumor)
  * Max Diameter group 1: >0 to ≤1.5 cm (cumulative if multiple residual lesions)
  * Max Diameter group 2: >1.5 cm (cumulative if multiple residual lesions)
OS with respect to MGMT promoter methylation status | 24 Months
  OS in patients with promoter methylation vs. no promoter methylation
PFS with respect to MGMT promoter methylation status | 24 Months
  PFS in patients with promoter methylation vs. no promoter methylation; determined according to modified RANO criteria and serial perfusion imaging
Quality of Life (QoL) questionnaire | 24 Months
  Assessed by European Organization for Research and Treatment (EORTC)- Quality of Life Questionnaires (QLQ C30/BN20)
Activities of daily living (ADL), assessed using the Barthel Index (Mahoney & Barthel, 1965). | 24 Months
  Change in functional outcomes as measured by BI from its baseline value.
Radiation-related (acute / early delayed / late) neurotoxicity | 24 Months
  Assessed by regular neurological examinations and serial MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Giordano, MD, Principal Investigator — Department of Radiation Oncology, University Medical Center Mannheim, University of Heidelberg, Germany; Kevin Petrecca, MD, Principal Investigator — Department of Neurosurgery, Montréal Neurological, Institute and Hospital, Montréal, Canada
Locations (19):
- United States (5):
  - Barrow Neurological Institute (SJHMC), Phoenix, Arizona
  - Stritch School of Medicine Loyola University, Maywood, Illinois
  - Long Island Jewish Medical Center, North Shore University Hospital, Lake Success, New York
  - Lenox Hill Hospital, Hofstra Northwell School of Medicine, New York, New York
  - West Virginia University, Morgantown, West Virginia
- Hospital Alemão Oswaldo Cruz, São Paulo, Brazil
- Montreal Neurological Institute and Hospital, Montreal, Quebec, Canada
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
- Germany (7):
  - University Hospital Augsburg, Augsburg
  - Charité - Universitätsmedizin, Berlin
  - St. Georg Hospital, Leipzig
  - University Hospital Mannheim, Mannheim
  - Technical University of Munich (TUM), Department of Radiation Oncology, Munich
  - Klinikum Stuttgart, Stuttgart
  - Helios University Hospital Wuppertal, Wuppertal
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea
- Spain (2):
  - Catalan Institute of Oncology (ICO), Barcelona
  - Hospital Reina Sofia, Córdoba
- The London Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giordano FA, Brehmer S, Abo-Madyan Y, Welzel G, Sperk E, Keller A, Schneider F, Clausen S, Herskind C, Schmiedek P, Wenz F. INTRAGO: intraoperative radiotherapy in glioblastoma multiforme-a phase I/II dose escalation study. BMC Cancer. 2014 Dec 22;14:992. doi: 10.1186/1471-2407-14-992. PMID 25535398
- [Background] Sarria GR, Sperk E, Han X, Sarria GJ, Wenz F, Brehmer S, Fu B, Min S, Zhang H, Qin S, Qiu X, Hanggi D, Abo-Madyan Y, Martinez D, Cabrera C, Giordano FA. Intraoperative radiotherapy for glioblastoma: an international pooled analysis. Radiother Oncol. 2020 Jan;142:162-167. doi: 10.1016/j.radonc.2019.09.023. Epub 2019 Oct 16. PMID 31629553
- [Background] Ayala Alvarez DS, Watson PGF, Popovic M, Heng VJ, Evans MDC, Panet-Raymond V, Seuntjens J. Evaluation of Dosimetry Formalisms in Intraoperative Radiation Therapy of Glioblastoma. Int J Radiat Oncol Biol Phys. 2023 Nov 1;117(3):763-773. doi: 10.1016/j.ijrobp.2023.04.031. Epub 2023 May 5. PMID 37150259
- [Background] Cifarelli CP, Jacobson GM. Intraoperative Radiotherapy in Brain Malignancies: Indications and Outcomes in Primary and Metastatic Brain Tumors. Front Oncol. 2021 Nov 11;11:768168. doi: 10.3389/fonc.2021.768168. eCollection 2021. PMID 34858846
- [Background] Sarria GR, Smalec Z, Muedder T, Holz JA, Scafa D, Koch D, Garbe S, Schneider M, Hamed M, Vatter H, Herrlinger U, Giordano FA, Schmeel LC. Dosimetric Comparison of Upfront Boosting With Stereotactic Radiosurgery Versus Intraoperative Radiotherapy for Glioblastoma. Front Oncol. 2021 Oct 28;11:759873. doi: 10.3389/fonc.2021.759873. eCollection 2021. PMID 34778080
- [Derived] Giordano FA, Brehmer S, Murle B, Welzel G, Sperk E, Keller A, Abo-Madyan Y, Scherzinger E, Clausen S, Schneider F, Herskind C, Glas M, Seiz-Rosenhagen M, Groden C, Hanggi D, Schmiedek P, Emami B, Souhami L, Petrecca K, Wenz F. Intraoperative Radiotherapy in Newly Diagnosed Glioblastoma (INTRAGO): An Open-Label, Dose-Escalation Phase I/II Trial. Neurosurgery. 2019 Jan 1;84(1):41-49. doi: 10.1093/neuros/nyy018. PMID 29528443